CLINICAL TRIAL: NCT00432419
Title: Therapeutic Intensification for HIV-associated Non-Hodgkin's Lymphoma by Autologous Transplantation of Either Unselected or CD34+-Selected Peripheral Blood Stem Cells, in Patients in First or Second Complete Remission. ANRS 131
Brief Title: Therapeutic Intensification of HIV-associated Non-Hodgkin's Lymphoma by Peripheral Blood Cell Transplantation Following Chemotherapy.
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: only one patient enrolled
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS131
Record Dates: First submitted 2007-02-05; First posted 2007-02-07 (Estimated); Last update posted 2011-12-22 (Estimated); Status verified 2011-12

CONDITIONS: HIV Infections; Lymphoma, Non-Hodgkin
Keywords: HIV; Non-Hodgkin's lymphoma; Peripheral blood stem cells transplantation
MeSH Terms: conditions — HIV Infections; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: autologous peripheral blood cell transplantation

SUMMARY:
Given the poor prognosis of HIV-associated non-Hodgkin's lymphoma (NHL) and it's still high incidence in HAART era, more intensive therapy is required in patients with initially severe stage of NHL or relapsing after first-line chemotherapy.

The purpose of this study is to evaluate the safety of an intensive chemotherapy followed by peripheral blood cell transplantation in these patients.

DETAILED DESCRIPTION:
Highly active antiretroviral therapy (HAART) has dramatically reduced mortality and morbidity of HIV-infected patients by decreasing the incidence of opportunistic infections and HIV-related malignancies such as Kaposi sarcoma. However, the frequency of NHL remains increased in these patients. Moreover, their prognostic remains poor comparing to HIV negative patients. This is mainly due to the type of NHL (aggressive B, and frequent stage IV) but also host factors such as immunodeficiency, co-infections (EBV, HHV8), and chemotherapy-HAART interactions. In the lack of new and significantly more efficient treatments, therapeutic intensification such as high-dose chemotherapy followed by autologous peripheral blood stem cell transplantation (ASCT), already tested in relapsed or partially responding HIV negative patients, could be an option in HAART controlled HIV+ patients with NHL, rather in first complete remission (CR) but with initially high International Prognosis Index (IPI above or equal to 2), or in second CR, whatever initial IPI. Positive selection CD34+ cells is an approach for depleting grafts of tumour cells and HIV DNA. However the delayed lymphocyte recovery following this process, may lead to increased incidence of opportunistic infections (OI) in HIV-infected patients. OI prophylaxis will be systematically associated.

Eligible patients will have peripheral blood stem cell (PBSC) mobilization and divided in two subgroups. Group A with 3-6 x 106 PBSC will not undergo CD34+ selection process and group B with more than 6 x 106 will undergo this process. The myeloablative conditioning process is the same in the two groups with total body irradiation before reinfusion of grafts.

Patients will be followed from week2 (W2) up to W60 with clinical and biological evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between 18 and 55 years old at screening
* Documented HIV-1 infection
* Currently HAART-treated
* Plasma HIV-RNA below 50 copies/ml at screening
* Lymphocyte T CD4+ count above or equal to 100/mm3 at the NHL diagnosis
* Histologically proven large cell NHL in first remission with classical poor prognostic factors (IPI above or equal to 2) or in second remission whatever IPI.
* Biological criteria of eligibility for intensive therapeutic
* Signed written informed consent
* Patient protected by the social security of one of the European community countries.

Exclusion Criteria:

* Burkitt NHL
* Central nervous system NHL
* Patients already treated by ASCT
* Ongoing infectious disease
* Psychiatric disease
* Left ventricular ejection fraction < 25%
* Creatinine clearance < 50 ml/min
* Hepatic failure
* Uncontrolled high blood pressure
* Chronic hepatitis C or B
* Participating in other trials.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2007-02; Primary Completion 2008-07 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Safety criteria defined as the occurrence of grades 3 or 4 adverse events in the 6 months following transplantation.

SECONDARY OUTCOMES:
Evaluation of:
HIV RNA
HIV DNA
Percentage and absolute count of CD3, CD4+ and CD8+ lymphocytes
Lymphocyte phenotypes and functions
TREC analysis
Immune reconstitution in vivo
Duration of aplasia

CONTACTS AND LOCATIONS:
Overall Officials: Yves LEVY, MD, PhD, Principal Investigator — Service d'Immunologie Clinique, Henri Mondor Hospital 94010 Creteil Cedex; Genevieve CHENE, MD, PhD, Study Director — INSERM Unit 593, Bordeaux
Locations (1):
- Servide d'Immunologie Clinique, Créteil, France